CLINICAL TRIAL: NCT07038967
Title: Assessment of Non-Center Involving Diabetic Macular Edema Progression in Early Postoperative Period After Phacoemulsification
Brief Title: Non-Center Involving Diabetic Macular Edema Progression in Early Postoperative Period After Phacoemulsification
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hatem Fawzy Abd Elfatah Abo saif, Lecturer of Ophthalmology, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: FMASU R127/2025
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Non-Center; Diabetic Macular Edema; Phacoemulsification
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with Grade I - Grade II nuclear cataract and non-center-involving diabetic macular edema (NCIDME)
  Interventions: Other: Coloured photography; Other: Fluorescein angiography; Other: Optical coherence tomography

INTERVENTIONS:
Other: Coloured photography — Coloured photography will be performed preoperatively and at 3 and 6 months postoperatively.
Other: Fluorescein angiography — Fluorescein angiography will be performed preoperatively and at 3 and 6 months postoperatively. The following features will be recorded on each angiography:
Other: Optical coherence tomography — Optical coherence tomography (OCT) scanning will be performed using the optical coherence tomography scanner OCT (OPTOVUE OCT). OCT will be performed preoperatively and at 3 and 6 months postoperatively.

SUMMARY:
This study aims to evaluate the progression of non-center-involving diabetic macular edema in the early postoperative period following phacoemulsification.

DETAILED DESCRIPTION:
Diabetic patients have been reported to have a higher prevalence of cataract and develop it at an earlier age compared with nondiabetic individuals.

According to recent population-based studies, diabetic macular edema (DME) is the most common cause of vision loss, with the incidence of non-center-involving DME (NCIDME) being higher than that of center-involving DME (CIDME). The prevalence of NCIDME in an urban south Indian population is 10.8%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sexes.
* Patients with Grade I - Grade II nuclear cataract and non-center-involving diabetic macular edema (NCIDME).

Exclusion Criteria:

* Traumatic cataract.
* Severe Non-Proliferative/ Proliferative Diabetic Retinopathy.
* Marked Asymmetry of retinopathy between both eyes.
* Mature senile cataract or severe lens opacity.
* Potentiality to have Phacotrabeculectomy surgery.
* Complications during or after the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will be conducted on 50 diabetic patients aged ≥18 years, both sexes, with Grade I - Grade II nuclear cataract and non-center-involving diabetic macular edema (NCIDME).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 6 months post-procedure
  Best Corrected Visual Acuity (BCVA) will be recorded.

SECONDARY OUTCOMES:
Intra ocular pressure | 6 months post-procedure
  Intra ocular pressure (IOP) will be recorded.
Central macular thickness (CMT) | 6 months post-procedure
  Central macular thickness (CMT) will be recorded.
Frequency distribution of Fluorescein leakage | 6 months post-procedure
  Frequency distribution of Fluorescein leakage will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.